CLINICAL TRIAL: NCT02496364
Title: Topical and Intravenous Use of Tranexamic Acid in Posterior Lumbar Interbody Fusion - A Prospective, Double-blind, Randomized Study
Brief Title: Evaluation of Topical and Intravenous Tranexamic Acid in Surgical Treatment of Lumbar Degenerative Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Dismissal from the institution
Sponsor: Vinicius Magno da Rocha, MD, MSc (Other Government)
Responsible Party: Sponsor-Investigator, Vinicius Magno da Rocha, MD, MSc, MD, Instituto Nacional de Traumatologia e Ortopedia
Organization: Instituto Nacional de Traumatologia e Ortopedia (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-2015
Record Dates: First submitted 2015-06-28; First posted 2015-07-14 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Lumbar Disc Degeneration; Surgical Procedure, Unspecified
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Observation (Other): Clinical data analysis
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
Evaluation of Topical and Intravenous Tranexamic Acid in Surgical Treatment of Lumbar Degenerative Disease

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Observation | 1